CLINICAL TRIAL: NCT03199963
Title: A Randomized, Double-blind, Placebo Controlled Trial of 4-Hydroxytamoxifen Gel for Reducing Breast Tissue Density in Women With BI-RADS Breast Density Categories C or D
Brief Title: Trial of 4-Hydroxytamoxifen (4-OHT) Gel in Women Aimed at Reducing Dense Breast Tissue
Acronym: 4WARD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Administrative - change in development strategy
Sponsor: BHR Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHR-700-301
Record Dates: First submitted 2017-06-21; First posted 2017-06-27 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-06

CONDITIONS: Mammographic Breast Density
Keywords: Mammographic; Breast; Density; BIRADS C or D
MeSH Terms: interventions — 4,17 beta-dihydroxy-4-androstene-3-one

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BHR-700 (0.2% 4-OHT gel) (Experimental): The gel formulation contains 2 mg/mL 4-OH tamoxifen (0.2%) in a clear, colorless, absorptive hydro-alcoholic gel base formulated to provide continuous release of 4-OH tamoxifen. A total of 8 mg/day (4 mg/breast) of 4-OH tamoxifen will be administered daily for 52 weeks.
  Interventions: Drug: 4-OH tamoxifen
- Matching Placebo Gel (Placebo Comparator): An absorptive hydroalcoholic gel preparation of the same ingredients as BHR-700, but without 4-OHT.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4-OH tamoxifen — 4-Hydroxytamoxifen (afimoxifene) gel
  Other Names: 4-OHT
  Arms: BHR-700 (0.2% 4-OHT gel)
Drug: Placebo — An absorptive hydroalcoholic gel preparation of the same ingredients as BHR-700, but without 4-OHT.
  Arms: Matching Placebo Gel

SUMMARY:
A study to determine the efficacy of 8 mg/day (4 mg/breast) of BHR-700 gel compared to placebo for reducing breast tissue density in women identified as having dense breast tissue upon analysis of screening mammography. The Primary Study Endpoint being the percent reduction of mammographic breast tissue density on a follow-up mammogram compared to the baseline mammogram after 52 weeks of treatment.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo-controlled study. Subjects will have been assessed as having mammographically dense breast (heterogeneously dense (C) or extremely dense (D), based on the American College of Radiology (ACR) Breast Imaging-Reporting and Data System (BIRADS©) fifth edition classification) for eligibility.

Approximately 330 subjects will be enrolled at approximately 25 sites in the US and the European Union. Subjects who give informed consent will be stratified, based on whether they are pre/peri or post-menopausal and randomized 2:1 within those groups to receive either 8 mg/day (4 mg/breast) 4-OHT or matching placebo for up to 52 weeks.

Subjects will apply the investigational gel to both breasts once per day until they have completed 52 weeks of study drug administration. There will be, in addition, an optional 52 weeks of open-label treatment for those subjects who choose to continue treatment. Subjects will capture daily gel administration in a diary to monitor compliance.

While on treatment, subjects will return to the clinic for study assessments, a review of adverse events (AEs) and to re-supply study gel at 13, 26, 39, weeks and at 52 weeks for those subjects who have agreed to take part in the open-label phase of the study. During the study, in a case of significant changes in bleeding pattern or other signs/symptoms which could be related to endometrial pathology, the Investigator will perform a uterine ultrasound followed by an endometrial biopsy if indicated.

Open-Label Treatment Phase

Secondary Outcome Measures: • Comparison of breast density measurements (Cumulus and Volpara) • Laboratory parameters will be summarized in a descriptive fashion. • Incidence and severity of AEs will be compared between BHR-700 gel and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women age 35 - 75 years with either heterogeneously dense (C) or extremely dense (D), breast tissue on 2D mammography, based on American College of Radiology (ACR) Breast Imaging-Reporting and Data System (BI-RADS©) fifth edition classification) in either breast within 3 months prior to randomization. Mammogram with BI-RADS final assessment category 1 or 2 (negative or benign findings).
2. If the participant is of childbearing potential, she must have a documented negative urine pregnancy test at the time of screening and randomization and no plans to become pregnant for the duration of study participation.
3. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Participants may not be receiving treatment with any investigational drug or biologic within 30 days of randomization or at any time during the study.
2. Women with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Tamoxifen.
3. Pregnant women are excluded from this study because the effects of 4-OHT gel on the developing human fetus at the recommended dose and route are unknown.
4. Pregnancy (independent of outcome) and/or lactation within 1 year prior to the screening mammogram.
5. Women with previous history of cancer (including invasive or intra-ductal breast cancer) except for non-melanoma skin cancer.
6. Women who have had a prior mastectomy (unilateral or bilateral), segmental mastectomy, reduction mammoplasty or breast augmentation including implants.
7. Women with surgical breast biopsy(s) performed within 3 years or core biopsy(s) performed within 1 year prior to the screening mammogram.
8. Women with an abnormal mammogram (BI-RADS final assessment category 3-probably benign, 4-suspicious, or 5-malignant findings). Women with BI-RADS 0 assessment (needs additional imaging evaluation) that are subsequently found to have negative (BI-RADS 1) or benign findings (BI-RADS 2), are NOT excluded.
9. Women with only synthetic 2D mammograms generated from 3D (tomosynthesis) are excluded as breast density measurements are not yet validated for synthetic mammograms. Women with combination 2D+3D mammograms are not excluded.
10. Women with active liver disease or thromboembolic disorder.
11. Women with skin conditions such as psoriasis, fungal infections, keloids etc., or tattoos and/or piercings, which in the opinion of the Investigator, would interfere with absorption of the Investigational Product.
12. Women who have had an abnormal gynecology exam within the last three years with clinically significant findings, such as secondary dysmenorrhea, polyps, or atypia, which in the opinion of the Investigator would interfere with the study.
13. Women who have received treatment with Selective Estrogen Receptor Modulators (SERMs) (e.g. tamoxifen, raloxifene) or aromatase inhibitors
14. Women taking estrogen containing contraceptives or Hormone Replacement Therapy (HRT) must discontinue the treatment a minimum of 6 months prior to the screening mammogram. Progestin only contraceptives are permitted.
15. Women with a concurrent illness, disease or condition that, in the opinion of the Investigator, would limit their compliance with study requirements or place them at additional risk.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — BHR Pharma, LLC
Locations (19):
- United States (17):
  - Mesa Obstetricians and Gynecologists/Cactus Clinical Research, Mesa, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - United Clinical Research, Beverly Hills, California
  - City of Hope, Duarte, California
  - USC-Keck Medical Center, Los Angeles, California
  - South Florida Medical Research, Aventura, Florida
  - Lake OB-GYN Associates of Mid-Florida, Leesburg, Florida
  - Physician Care Clinical Research, LLC, Sarasota, Florida
  - Affiliated Clinical Research, Inc., Las Vegas, Nevada
  - Center for Women's Health and Wellness, Plainsboro, New Jersey
  - Bosque Women Care/Cactus Clinical Research, Albuquerque, New Mexico
  - Carolina Women's Research and Wellness Center, Durham, North Carolina
  - Aventiv Research, Inc., Columbus, Ohio
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - University of Virginia Medical Park Northridge, Charlottesville, Virginia
  - Overlake Internal Medicine Associates, PS, Bellevue, Washington
  - Dedicated Women's Health Specialists, Puyallup, Washington
- Private Practice - Gynecology, Frankfurt am Main, Hesse, Germany
- Instituto Palacios Salud de La Mujer, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Blinded Phase - Overall Study
Arm/Group | BHR-700 (0.2% 4-OHT Gel) | Matching Placebo Gel
Started | 149 | 74
Received at Least 1 Gel Application | 149 | 73
Completed (Completed 52 week visit) | 16 | 8
Not Completed | 133 | 66
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Lost to Follow-up | 9 | 2
Not completed — Adverse Event | 10 | 5
Not completed — Study was terminated early by the Sponsor for administrative reasons. | 109 | 54
Period: Optional Open-Label Phase - BHR-700
Arm/Group | BHR-700 (0.2% 4-OHT Gel) | Matching Placebo Gel
Started | 7 | 6
Completed | 0 | 0
Not Completed | 7 | 6
Not completed — Study terminated early by Sponsor for administrative reasons; data contribution was negligible. | 7 | 5
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 223 subjects were enrolled in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | BHR-700 (0.2% 4-OHT Gel) | Matching Placebo Gel | Total
Number analyzed (Participants) | 149 | 74 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (9.23) | 56.2 (9.63) | 54.9 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 74 | 223
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 7 | 18
  White | 132 | 65 | 197
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 140 | 71 | 211
  Germany | 3 | 1 | 4
  Spain | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Percent Reduction of Mammographic Dense Breast (MBD) Tissue on a Follow-up Mammogram Compared to the Baseline Mammogram After 52 Weeks of Treatment.
Description: Percent MBD at screening compared to percent MBD after 52 weeks of treatment with either BHR-700 or Placebo.
Time Frame: Blinded Phase: Baseline; Week 52
Population: Study was terminated early for administrative and not safety reasons; an abbreviated clinical study report was prepared and results were limited to safety parameters only. This outcome was not collected and therefore cannot be reported.
Arm/Group | BHR-700 (0.2% 4-OHT Gel) | Matching Placebo Gel
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number and Severity of Adverse Events (AEs)
Description: AEs monitored and reported throughout study
Time Frame: Blinded Phase: Baseline; Weeks 13, 26, 39, 52/EOS and Open Label Phase
Population: A total of 223 subjects were enrolled in this study; 222 subjects were randomized to the study treatment and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- BHR-700 (0.2% 4-OHT Gel) in Blinded Phase; Open Label BHR-700 (0.2% 4-OHT Gel) Following BHR-700 in Blinded Phase; Open Label BHR-700 (0.2% 4-OHT Gel) Following Placebo in Blinded Phase: The gel formulation contains 2 mg/mL 4-OH tamoxifen (0.2%) in a clear, colorless, absorptive hydro-alcoholic gel base formulated to provide continuous release of 4-OH tamoxifen. A total of 8 mg/day (4 mg/breast) of 4-OH tamoxifen will be administered daily for 52 weeks.
  4-OH tamoxifen: 4-Hydroxytamoxifen (afimoxifene) gel
- Matching Placebo Gel in Blinded Phase: An absorptive hydroalcoholic gel preparation of the same ingredients as BHR-700, but without 4-OHT.
  Placebo: An absorptive hydroalcoholic gel preparation of the same ingredients as BHR-700, but without 4-OHT.
Arm/Group | BHR-700 (0.2% 4-OHT Gel) in Blinded Phase | Matching Placebo Gel in Blinded Phase | Open Label BHR-700 (0.2% 4-OHT Gel) Following BHR-700 in Blinded Phase | Open Label BHR-700 (0.2% 4-OHT Gel) Following Placebo in Blinded Phase
Number analyzed (Participants) | 149 | 73 | 7 | 6
Participants
  Subjects with at least one mild AE | 56 | 31 | 2 | 1
  Subjects with at least one moderate AE | 49 | 29 | 2 | 1
  Subjects with at least one severe AE | 8 | 4 | 1 | 0

3. Secondary Outcome: Change in Serum Concentration of Sex Hormone Binding Globulin (SHBG) From Baseline to Week 52/End of Study (EOS)
Description: SHBG levels at baseline will be compared to levels at Week 52/EOS
Time Frame: Blinded Phase: Baseline; Week 52/EOS
Population: This parameter captures data from Week 52 or End of Study for subjects who stopped treatment at various timepoints before the 52 weeks.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | BHR-700 (0.2% 4-OHT Gel) | Matching Placebo Gel
Number analyzed (Participants) | 111 | 56
mg/L | 0.1 (1.6) | 0.3 (1.6)

4. Secondary Outcome: Change in Serum Concentration of: Cholesterol, Triglycerides, High-density Lipoprotein (HDL), and Low-density Lipoprotein (LDL).
Description: Lipid levels at baseline will be compared to levels measured at time-points in the study
Time Frame: Blinded Phase: Baseline; Weeks 26, 52/EOS.
Population: Study was terminated early for administrative and not safety reasons; an abbreviated clinical study report was prepared and results were limited to safety and pharmacokinetic (PK)/pharmacodynamic (PD) parameters only. Of all subjects that attended the Week 52/End of Study visit, only 24 subjects completed 52 weeks of treatment. All other subjects stopped treatment at various timepoints before the 52 weeks.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | BHR-700 (0.2% 4-OHT Gel) | Matching Placebo Gel
Number analyzed (Participants) | 148 | 73
mmol/L
  Cholesterol (mmol/L) - Change from Baseline to Week 26: number analyzed (Participants) | 59 | 33
  Cholesterol (mmol/L) - Change from Baseline to Week 26 | -0.1 (0.6) | -0.2 (0.7)
  Cholesterol (mmol/L) - Change from Baseline to Week 52/EOS: number analyzed (Participants) | 116 | 58
  Cholesterol (mmol/L) - Change from Baseline to Week 52/EOS | 0.1 (0.7) | 0.0 (0.7)
  Triglycerides (mmol/L) - Change from Baseline to Week 26: number analyzed (Participants) | 59 | 33
  Triglycerides (mmol/L) - Change from Baseline to Week 26 | -0.2 (1.2) | -0.2 (0.6)
  Triglycerides (mmol/L) - Change from Baseline to Week 52/EOS: number analyzed (Participants) | 116 | 58
  Triglycerides (mmol/L) - Change from Baseline to Week 52/EOS | -0.1 (0.8) | 0.0 (0.8)
  HDL Cholesterol (mmol/L) - Change from Baseline to Week 26: number analyzed (Participants) | 59 | 33
  HDL Cholesterol (mmol/L) - Change from Baseline to Week 26 | -0.0 (0.3) | 0.0 (0.2)
  HDL Cholesterol (mmol/L) - Change from Baseline to Week 52/EOS: number analyzed (Participants) | 116 | 58
  HDL Cholesterol (mmol/L) - Change from Baseline to Week 52/EOS | 0.0 (0.2) | 0.0 (0.3)
  LDL Cholesterol (mmol/L) - Change from Baseline to Week 26: number analyzed (Participants) | 59 | 33
  LDL Cholesterol (mmol/L) - Change from Baseline to Week 26 | 0.0 (0.6) | -0.1 (0.7)
  LDL Cholesterol (mmol/L) - Change from Baseline to Week 52/EOS: number analyzed (Participants) | 116 | 56
  LDL Cholesterol (mmol/L) - Change from Baseline to Week 52/EOS | 0.1 (0.5) | -0.0 (0.7)

5. Secondary Outcome: Change in Serum Concentration of Select Bone Biomarkers: Bone Specific Alkaline Phosphatase (BSAP) (U/L)
Description: Bone biomarker levels (BSAP) at baseline will be compared to levels measured at Week 52.
Time Frame: Blinded Phase: Baseline; Week 52/EOS
Population: 133 participants in the BHR-700 arm and 65 in the placebo arm were included at baseline. Data from 97 BHR-700 and 48 placebo participants are reported at Week 52/EOS.
Measure: Mean (Standard Deviation); unit: BSAP in U/L
Arm/Group | BHR-700 (0.2% 4-OHT Gel) | Matching Placebo Gel
Number analyzed (Participants) | 97 | 48
BSAP in U/L | 1.0 (4.1) | 0.7 (3.3)

6. Secondary Outcome: Number of Participants With Measurable Plasma Concentrations of the E and Z Isomers of 4-OHT by Visit
Description: Blood samples will be taken to measure plasma concentrations of 4-OHT at time-points in the study
Time Frame: Blinded Phase: Weeks 13, 26, 52/EOS
Population: Concentrations measured only in participants who received BHR-700. Of all subjects that attended the Week 52/End of Study visit, only 24 subjects completed 52 weeks of treatment. All other subjects stopped treatment at various timepoints before the 52 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | BHR-700 (0.2% 4-OHT Gel) | Matching Placebo Gel
Number analyzed (Participants) | 179 | 0
Participants
  Week 13 E-4-OHT: number analyzed (Participants) | 140 | 0
  Week 13 E-4-OHT: Participants with measurable concentration | 12 |
  Week 13 E-4-OHT: Participants with concentration below lower limit of quantitation | 128 |
  Week 26 E-4-OHT: number analyzed (Participants) | 95 | 0
  Week 26 E-4-OHT: Participants with measurable concentration | 7 |
  Week 26 E-4-OHT: Participants with concentration below lower limit of quantitation | 88 |
  Week 52/EOS E-4-OHT: Participants with measurable concentration | 0 |
  Week 52/EOS E-4-OHT: Participants with concentration below lower limit of quantitation | 179 |
  Week 13 Z-4-OHT: number analyzed (Participants) | 140 | 0
  Week 13 Z-4-OHT: Participants with measurable concentration | 75 |
  Week 13 Z-4-OHT: Participants with concentration below lower limit of quantitation | 65 |
  Week 26 Z-4-OHT: number analyzed (Participants) | 95 | 0
  Week 26 Z-4-OHT: Participants with measurable concentration | 48 |
  Week 26 Z-4-OHT: Participants with concentration below lower limit of quantitation | 47 |
  Week 52/EOS Z-4-OHT: Participants with measurable concentration | 16 |
  Week 52/EOS Z-4-OHT: Participants with concentration below lower limit of quantitation | 163 |

7. Secondary Outcome: Change in Serum Concentration of Select Bone Biomarkers:Type I Collagen C-Telopeptides (CTx) (pg/mL)
Description: Bone biomarker levels (CTx) at baseline will be compared to levels measured at Week 52.
Time Frame: Blinded Phase: Baseline; Week 52/EOS
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | BHR-700 (0.2% 4-OHT Gel) | Matching Placebo Gel
Number analyzed (Participants) | 97 | 48
pg/mL | -19.6 (162) | 3.7 (155.5)

ADVERSE EVENTS:
Time Frame: Blinded and Open Label Portions of the Study up to 104 Weeks
Description: The Safety Population is the population of all patients who receive at least 1 dose of study treatment.
Arm/Group | BHR-700 (0.2% 4-OHT Gel) in Blinded Phase | Matching Placebo Gel in Blinded Phase | Open Label BHR-700 (0.2% 4-OHT Gel) Following BHR-700 in Blinded Phase | Open Label BHR-700 (0.2% 4-OHT Gel) Following Placebo in Blinded Phase
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/73 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/149 | 0/73 | 1/7 | 0/6
Other Adverse Events (participants affected / at risk) | 71/149 | 43/73 | 3/7 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BHR-700 (0.2% 4-OHT Gel) in Blinded Phase (N=149) | Matching Placebo Gel in Blinded Phase (N=73) | Open Label BHR-700 (0.2% 4-OHT Gel) Following BHR-700 in Blinded Phase (N=7) | Open Label BHR-700 (0.2% 4-OHT Gel) Following Placebo in Blinded Phase (N=6)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BHR-700 (0.2% 4-OHT Gel) in Blinded Phase (N=149) | Matching Placebo Gel in Blinded Phase (N=73) | Open Label BHR-700 (0.2% 4-OHT Gel) Following BHR-700 in Blinded Phase (N=7) | Open Label BHR-700 (0.2% 4-OHT Gel) Following Placebo in Blinded Phase (N=6)
Nasopharyngitis (Infections and infestations) | 12 | 5 | 0 | 0
Sinusitis (Infections and infestations) | 9 | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 8 | 0 | 0
Urinary tract infection (Infections and infestations) | 6 | 3 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 5 | 1 | 0 | 0
Influenza (Infections and infestations) | 4 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0
Heliobacter infection (Infections and infestations) | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 1 | 0 | 0
Lip infection (Infections and infestations) | 1 | 0 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 2 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Peripheral arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 4 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 4 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 3 | 3 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 1 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast discoloration (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 2 | 0 | 0
Menstruation delayed (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Vaginal cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast calcifications (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Nipple disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal erosion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestinal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 4 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Acne cystic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 6 | 2 | 0 | 0
Pain (General disorders) | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Application site reaction (General disorders) | 1 | 0 | 0 | 0
Axillary pain (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Medical device site ulcer (General disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 7 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 5 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Musculoskeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Body temperature increased (Investigations) | 3 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 0 | 0
QRS axis abnormal (Investigations) | 1 | 0 | 0 | 0
Rheumatoid factor increased (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0
Mammogram abnormal (Investigations) | 0 | 1 | 0 | 0
Protein S decreased (Investigations) | 0 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 4 | 3 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 0 | 0
Libido increased (Psychiatric disorders) | 1 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 0 | 0
Ear pruritis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 2 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Product odour abnormal (Product Issues) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemangioma of the liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Dolichocolon (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2
Eye pain (Eye disorders) | 0 | 0 | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Other (Not Including Serious) Adverse Events entries are based on number of subject in the intention-to-treat (ITT) population (blinded phase, safety population). Includes all adverse events reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT03199963/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT03199963/SAP_001.pdf